CLINICAL TRIAL: NCT02973334
Title: Acute Effects of Artificial Sweeteners' or Sugar's Ingestion on Hemodynamic and Metabolic Stress Response: An Exploratory, Randomized, Cross-over Trial in Healthy Young Women.
Brief Title: Acute Effects of Artificial Sweeteners or Sugar on Hemodynamic and Metabolic Stress Responses
Acronym: EduStress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Full Professor, University of Lausanne
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 316/15
Record Dates: First submitted 2016-11-14; First posted 2016-11-25 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Normal Subjects
Keywords: sweeteners; sugar; stress response
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sugar (Experimental): Effects of ingestion of sugar-sweetened beverages on acute stress response
  Interventions: Other: Ingestion of sugar-sweetened beverages
- Artificial sweetener (Experimental): Effects of ingestion of artificially-sweetened beverages on acute stress response
  Interventions: Other: Ingestion of artificially-sweetened beverages
- Water (Active Comparator): Effects of ingestion of water on acute stress response
  Interventions: Other: Ingestion of water

INTERVENTIONS:
Other: Ingestion of artificially-sweetened beverages — From t=60 to the end of the metabolic test, volunteers will ingest 7 beverages containing non nutritive sweeteners (25 mL / beverage) every 15 minutes after 10-sec mouth rinsing.
  Arms: Artificial sweetener
Other: Ingestion of sugar-sweetened beverages — From t=60 to the end of the metabolic test, volunteers will ingest 7 beverages containing sugar (25 mL / beverage) every 15 minutes after 10-sec mouth rinsing.
  Arms: Sugar
Other: Ingestion of water — From t=60 to the end of the metabolic test, volunteers will ingest 7 water beverages (25 mL / beverage) every 15 minutes after 10-sec mouth rinsing.
  Arms: Water

SUMMARY:
This exploratory study aims at investigating the acute effects of artificially sweetened and sugar beverage consumption (as compared to water consumption) on acute hemodynamic and metabolic stress response.

DETAILED DESCRIPTION:
This single-center study included five visits. The first two visits (screening and familiarization) allowed checking the eligibility of the volunteers. In case of inclusion, the subjects were assigned to a sequence of three experimental conditions (water, sugar and artificial sweeteners), in a randomized, crossover design.

The experimental test was divided into 5 stages:

1. a 90 minutes baseline period (t=0-90 min),
2. a 30-min mental stress (MS; t=90-120 min), consisting in 5-min periods of Stroop's color word conflict test alternated with 5-min periods of mental arithmetic test.
3. a 30-min MS recovery period (t=120-150),
4. a 3-min cold pressure test (CPT) was carried out, aiming at immersing one volunteer's forearm in an ice water container at 3°C,

3) a 15-min CPT recovery period (t=120-150). 60 min after the beginning of the metabolic test, volunteers will drink 25 mL every 15 min, after 10-sec mouth rinsing, of either an artificially- or sugar-sweetened beverages or water (control).

Hemodynamic stress responses will be measured by repeated blood pressure, heart rate and cardiac output. Repeated venous blood samples will allow to assess metabolic stress responses.

Each condition (water, artificial sweeteners and sugar) will be preceded by a 2-day run-in period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Caucasian
* Normal Body Mass Index (18.5 ≤BMI≤ 25 kg/m2)
* Monophasic oral contraceptive

Exclusion Criteria:

* Hypertension (Blood pressure >140/90 mmHg)
* History or actual psychologic/cardiovascular troubles
* Anemia anamnesis
* Being Pregnant
* Weight < 50 kg
* Blood donation or participation to another study < 8 weeks
* Claustrophobia
* Consumption of sugar/artifically-sweetened beverages drinks > 5 dL/d
* Visual disturbances (daltonism)
* Low to moderate physical activity (> 4h/wk)
* Smoker and narcotic consumption
* Caffeine (> 400 mg/d) and/or alcohol (> 10g/d) consumption
* Medical treatment
* Weight variation > 3kg during the last month

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Hemodynamic changes | Differences observed between 90-min baseline and stress (30-min mental stress and 3-min cold pressure test)
  Hemodynamic changes elicited by stress will be assessed by means of systemic vascular resistance calculated as (blood flow):(mean arterial pressure, and expressed in arbitrary units

SECONDARY OUTCOMES:
Changes in concentration of blood glucose | Blood samples will be collected 30, 60, 75, 85, 95, 100, 110, 120, 125, 135, 145, 153, 158, and 163 minutes after the beginning of the test
  Blood glucose concentration will be measured in fasting conditions and during stress tests with the glucose oxidase method and expressed in mg/dl
Changes in concentration of blood insulin | Blood samples will be collected 30, 60, 75, 85, 95, 100, 110, 120, 125, 135, 145, 153, 158, and 163 minutes after the beginning of the test
  Blood insulin concentration will be measured by ELISA and expressed in mU/L
Changes in blood non-esterified fatty acid concentration | Blood samples will be collected 30, 60, 75, 85, 95, 100, 110, 120, 125, 135, 145, 153, 158, and 163 minutes after the beginning of the tes
  Blood non-esterified fatty acid concentration will be measured by a colorimetric method and expressed in mmol/L
Metabolic changes | Differences observed between 90-min baseline and stress (30-min mental stress and 3-min cold pressure test)
  Metabolic changes elicited by stress will be continually monitored from respiratory gas exchanges by indirect calorimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Luc TAPPY, Professor, Principal Investigator — Department of Physiology, University of Lausanne, Switzerland
Locations (1):
- University of Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No